CLINICAL TRIAL: NCT05282329
Title: Efficacy of Transcranial Alternating Current Stimulation (tACS) as an Add-on Treatment for Auditory Hallucinations in Refractory Schizophrenia: A Randomized, Double-blind, Sham-controlled Trial
Brief Title: Efficacy of tACS for Treatment of Auditory Hallucinations in Refractory Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tACS-TJAH
Record Dates: First submitted 2022-02-14; First posted 2022-03-16 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tACS group (Experimental): Participants receive tACS 20-min sessions in a 5-day sequence for four consecutive weeks,combined with original and stable medication. Active group participants were administered 2 mA alternating current delivered with gamma frequency, delivered over the temporal lobe.
  Interventions: Device: Transcranial alternating Current Stimulation (tACS)-active
- Sham group (Sham Comparator): Controls received sham stimulation with the same protocol.
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)-sham

INTERVENTIONS:
Device: Transcranial alternating Current Stimulation (tACS)-active — Transcranial alternating current stimulation (tACS) employs a weak electric current for non-invasive brain stimulation with a sine-wave waveform, targeting brain oscillations in a frequency-specific manner. daily tACS sessions were scheduled in a 5-day sequence for four consecutive weeks, and each session lasted 20minutes. Participants were administered 2 mA alternating current delivered with gamma frequency, delivered over the temporal lobe.
  Arms: tACS group
Device: Transcranial Alternating Current Stimulation (tACS)-sham — Transcranial alternating current stimulation (tACS) employs a weak electric current for non-invasive brain stimulation with a sine-wave waveform, targeting brain oscillations in a frequency-specific manner. Controls received sham stimulations with the same protocol.
  Arms: Sham group

SUMMARY:
The aim of this study is to evaluate the feasibility and efficacy of transcranial alternating current stimulation (tACS) as an add-on treatment for auditory hallucinations in refractory schizophrenia. Meanwhile, we aim to evaluate the effect of tACS on cognitive function of schizophrenia patients. we hypothesize tACS would improve refractory auditory hallucination symptoms in schizophrenia by regulating the gamma frequency band of temporal lobe。

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled study to detect the effect of tACS for treatment of refractory auditory hallucinations in schizophrenia. 50 participants were randomly assigned 1:1 to tACS group or sham-control group. For both active and sham group, daily tACS sessions were scheduled in a 5-day sequence for four consecutive weeks, and each session lasted 20minutes. Based on the original and stable medication, active participants were administered 2 mA alternating current delivered with gamma frequency, delivered over the temporal lobe, while controls received sham stimulations with the same protocol. Scale assessments are performed at baseline, week 2, week 4 and week 6. Collection of blood took place at baseline, week 4 and week 6.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants aged 18-70 with DSM-5-defined schizophrenia or schizophrenia-like disorder.
2. Duration of illness > 12 weeks.
3. Being clinically stable and on an adequate therapeutic dose of antipsychotics for at least 8 weeks prior to enrolment.
4. Junior high school education or above
5. After treatment with ≥ 2 different antipsychotics (greater than the equivalent dose of chlorpromazine 600mg), the curative effect was poor (CGI ≥ 4 points or the PANSS score reduction rate since this treatment was less than 20%)
6. Agreement to participate in the study and provide the written informed consent.

Exclusion Criteria:

1. Having unstable medical conditions, current psychiatric comorbidity or active substance use disorder (in exception to caffeine and/or tobacco)
2. Having Serious physical diseases or nervous system diseases;
3. Having any brain device / implant, including cochlear implant and aneurysm clip;
4. Having a history or family history of autoimmune diseases or immune diseases;
5. Pregnancy or breastfeeding at enrollment;
6. Skin lesions on scalp at the area of electrode application.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
The change over time in the score of Psychotic Symptom Rating Scales (PSYRATS) | baseline, week 2, week 4, week 6
  The main objective is to explore whether tACS combined with antipsychotics could improve refractory auditory hallucinations in schizophrenia after 4-week treatment. PSYRATS were assessed at baseline and week 2, 4, 6. Higher total score of the scale means more severe auditory hallucinations symptoms.

SECONDARY OUTCOMES:
The change over time in the score of Hamilton Depression Rating Scale (HAMD-17) | baseline, week 2, week 4, week 6
  The change over time in the score of Hamilton Depression Rating Scale (HAMD-17)The aim is to explore whether tACS combined with antipsychotics could alleviate the severity of depressive symptoms as measured with HAMD-17 in refractory schizophrenia after 4-week treatment. Hamilton Depression Rating Scale (HAMD-17) was used to evaluate the severity of symptoms of depression. Higher total score of the scale means more severe depressive symptoms.
The change over time in the score of Hamilton Anxiety Rating Scale (HAMA) | baseline, week 2, week 4, week 6
  The aim is to explore whether tACS combined with antipsychotics could alleviate the severity of anxious symptoms as measured with HAMA in refractory schizophrenia after 4-week treatment. Hamilton Anxiety Rating Scale (HAMA) was used to evaluate the severity of symptoms of anxiety. Higher total score of the scale means more severe anxious symptoms.
The change of scores in cognition | baseline, week 4
  The aim is to observe whether active-stimuli in addition to regular treatment with antipsychotics will improve the cognitive function as measured with the MATRICS Consensus Cognitive Battery after 4 weeks of treatment compared to sham-stimuli, and investigators assess the scale at baseline and week 4.
The changes of levels of Brain Derived Neurotrophic Factor in peripheral blood from baseline to week 6 | baseline, week 4, week 6
  The aim is to investigate the change of Brain Derived Neurotrophic Factor level in peripheral blood as active stimuli in addition to regular medical treatment after 4 weeks of treatment compared to sham stimuli, and EDTA tubes were used to collect 5ml of peripheral blood at baseline, weeks 4, and 6 before feeding. The plasma was extracted after centrifugation, and the concentration of BDNF in plasma was detected by ELISA.
The change of scores of Adverse events scale from baseline to week 4 | week 1, week 2, week 3, week 4
  The aim is to evaluate the adverse effects during the treatment.
The change of Gamma band activity before and after intervention | baseline, week4, week 6
  The aim is to observe the changes in gamma band activity before and after intervention. EEG signals were recorded at baseline, 4 and 6 weeks. Gamma has been interpreted as an imbalance between excitation and inhibition, and is significantly associated with positive symptoms in schizophrenia. Changes in Gamma PSD before and after intervention were calculated by resting state EEG. In addition, 40hz - auditory homeostasis was collected to calculate whether the power of auditory evoked potentials changed before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China